CLINICAL TRIAL: NCT03103594
Title: Comparison of the Treatment of Refractory Bladder Pain Syndrome With Dimethyl Sulfoxide (DMSO) Alone and DMSO as a Carrier Molecule for Botulinum Toxin A Instillation.
Brief Title: Comparison of the Treatment of Refractory Bladder Pain Syndrome With DMSO and DMSO With Botulinum Toxin A
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Society for Urodynamics and Female Urology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 821084
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Dimethyl Sulfoxide; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will not be notified of which arm they are randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DMSO alone (Active Comparator): Half of the patients will undergo DMSO instillation
  Interventions: Drug: DMSO
- DMSO with Botox (Experimental): The other half will be randomized to DMSO mixed with 200U of botulinum toxin instillation
  Interventions: Drug: DMSO; Drug: Botox

INTERVENTIONS:
Drug: DMSO — DMSO will be instilled intravesically.
Drug: Botox — Botox will be instilled intravesically with DMSO.
  Arms: DMSO with Botox

SUMMARY:
The purpose of this research study is to evaluate the efficacy of intravesical botulinum A toxin and DMSO in women with bladder pain syndrome who have not responded to first-line treatments. Bladder pain syndrome is suprapubic pain with bladder filling as well as frequency, urgency, and nocturia in the absence of urinary tract infection or other pathology. DMSO has been shown to reduce pain in women with bladder pain syndrome as well as increase bladder absorption of various drugs. Botulinum toxin A has also been shown to improve pain in women with bladder pain syndrome when injected into the bladder suburothelium via a cystoscope. The main objective of this study is to assess if DMSO can deliver botulinum toxin to the suburothelium of the bladder to produce the same effect as direct injection of Botulinum toxin and a better effect than DMSO alone.

DETAILED DESCRIPTION:
Bladder pain syndrome (BPS) is defined by the AUA as an unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than six weeks duration, in the absence of infection or other identifiable causes. If the patient also has atypical cystoscopic and histological features then they are categorized as having Interstitial Cystitis.

Dimethyl sulfoxide (DMSO) is an FDA-approved treatment for BPS and is thought to work by its exceptional solvent properties. It has been shown to desensitize nociceptive pathways in the lower urinary tract. It has been shown to improve pain in women with refractory BPS utilized initially in the 1960s when Stewart began instilling it intravesically.

DMSO has also long been known to increase absorption of other agents instilled into the bladder. In a Japanese study, female rats were instilled with a chemotherapeutic agent as well as DMSO or just the chemotherapy alone. Using fluorescence they were able to show that with DMSO the chemotherapy drug was able to extend into the deeper layers of the bladder wall compared to just the epithelial layer in those that received just the chemotherapy drug.

Botulinum toxin A is thought to work by decreasing acetylcholine release and causing paralysis of muscle tissue in smooth and striated muscle. It has been shown to improve pain in women with BPS when administered via injection It has also been shown to improve frequency/urgency in patients with BPS. Botulinum toxin has been shown to be effective when injected into the bladder urothelium for patients with overactive bladder.

The investigators hypothesize that DMSO can deliver botulinum toxin to the suburothelium of the bladder to produce the same or similar effect as direct injection. Prior studies in women with refractory OAB showed that instillation resulted in improved continence, urgency, and quality of life as measured by UDI-6 and IIQ-7 questionnaires. In a prospective randomized study patients who received bladder instillation of liposome encapsulated botulinum toxin had improvement of their overactive bladder symptoms.

The investigators hope to show this improvement in patients with bladder pain syndrome/interstitial cystitis. Botulinum toxin has a variable duration of effect in the bladder similar to other parts of the body. In one study, duration of improvement was estimated to be 7 to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 18-75 years, capable of giving consent
2. Previously diagnosed with bladder pain syndrome/Interstitial cystitis that is refractory to dietary and behavioral modifications with an O'Leary-Sant score of 12 at baseline.
3. Patients should have no change in their oral medications for bladder pain syndrome in the last 3 months
4. Patients with respiratory conditions will be required to present a medical clearance before administration Botulinum toxin.

Exclusion Criteria:

* 1. active treatment for bladder pain syndrome that is satisfactory to reduce symptoms 2. Urinary tract infection in the previous 6 weeks 3. History of bladder cancer, high grade dysplasia or radiation cystitis 4. Current or planned pregnancy in the next 6 months 5. Any change to regimen for lower urinary tract manipulations in the past 8 weeks (including Interstim, Tibial Nerve stimulation, pelvic floor muscle training, and biofeedback) 6. Previous botulinum toxin instilled or injected in the last 6 months. 7. Subjects cannot be homeless persons, or have active drug/alcohol dependence or abuse history 8. Subjects cannot have a personal history of a hypersensitivity reaction to Botulinum Toxin A

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pain Score | 6 months
  We hypothesize that DMSO can deliver botulinum toxin to the suburothelium of the bladder to produce the same effect as direct injection of botulinum toxin via cystoscopy. The primary endpoint will be a pain score as measured by visual analog scale at 2 months post-instillation compared to pre-instillation pain score. We hypothesize that the effect of DMSO will have dissipated by that point and any improvement in pain will be attributable to the effects of botox.

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Smith, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.

REFERENCES:
- [Background] D'Ascanio P, Pompeiano M, Tononi G. Inhibition of vestibulospinal reflexes during the episodes of postural atonia induced by unilateral lesion of the locus coeruleus in the decerebrate cat. Arch Ital Biol. 1989 Mar;127(2):81-97. PMID 2719523
- [Background] Cui Y, Zhou X, Zong H, Yan H, Zhang Y. The efficacy and safety of onabotulinumtoxinA in treating idiopathic OAB: A systematic review and meta-analysis. Neurourol Urodyn. 2015 Jun;34(5):413-9. doi: 10.1002/nau.22598. Epub 2014 Mar 28. PMID 24676791
- [Background] Lucioni A, Bales GT, Lotan TL, McGehee DS, Cook SP, Rapp DE. Botulinum toxin type A inhibits sensory neuropeptide release in rat bladder models of acute injury and chronic inflammation. BJU Int. 2008 Feb;101(3):366-70. doi: 10.1111/j.1464-410X.2007.07312.x. PMID 18184328
- [Background] Smith CP, Radziszewski P, Borkowski A, Somogyi GT, Boone TB, Chancellor MB. Botulinum toxin a has antinociceptive effects in treating interstitial cystitis. Urology. 2004 Nov;64(5):871-5; discussion 875. doi: 10.1016/j.urology.2004.06.073. PMID 15533466
- [Background] Birder LA, Kanai AJ, de Groat WC. DMSO: effect on bladder afferent neurons and nitric oxide release. J Urol. 1997 Nov;158(5):1989-95. doi: 10.1016/s0022-5347(01)64199-5. PMID 9334655
- [Background] Stewart BH, Branson AC, Hewitt CB, Kiser WS, Straffon RA. The treatment of patients with interstitial cystitis, with special reference to intravesical DMSO. Trans Am Assoc Genitourin Surg. 1971;63:69-74. No abstract available. PMID 5137793